CLINICAL TRIAL: NCT00141362
Title: An Open-Label, Extension Safety and Efficacy Study of Pregabalin in Patients With Chronic Neuropathic Pain.
Brief Title: Evaluate Long-Term Safety and Efficacy of Pregabalin in Patients With Chronic Neuropathic Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-000-166
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-01-01 (Estimated); Status verified 2006-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
Evaluate long-term safety and efficacy of pregabalin in patients with chronic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for the preceding double-blind BID study in diabetic neuropathy or postherpetic neuralgia.
* Must have received study medication under double-blind conditions.

Exclusion Criteria:

* Patients cannot participate if they experienced a serious adverse event during the previous double-blind BID study which was determined to be related to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325
Dates: Start 2001-10; Study Completion 2005-08

PRIMARY OUTCOMES:
Safety and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer